

# **Statistical Analysis Plan**

# **MoLiMoR**

<u>Mo</u>dulation of the FOLFIRI-based standard 1st-<u>li</u>ne therapy with cetuximab, controlled by <u>mo</u>nitoring the <u>R</u>AS mutation load by liquid biopsy in RAS-mutated MCRC patients

A randomized phase II study with FOLFIRI-based 1st-line therapy with or without intermittent cetuximab

**Study number:** 4213000 MoLiMoR-Study Phase II

Medication: Cetuximab

**Document ID:** MoLiMoR SAP v2.0 2024SEP13.docx

Version: Version v2.0

Date: 13SEP2024

**Sponsor:** TheraOP gGmbH

Represented by Hanno Härtlein

Winchesterstraße 3 D-35394 Gießen

Germany

Phone: +49 (0)641 / 94436-0 Fax: +49 (0)641 / 94436-70

Author: Alcedis GmbH, Winchesterstraße 3, D-35394

Gießen, Germany

Dr. Christine Windemuth-Kieselbach

Dr. Maximilian Parr

**Protocol (version, date):** Final (v3.0 including Amendment 1), 09MAR2021

### **MoLiMoR**

Modulation of the FOLFIRI-based standard 1st-line therapy with cetuximab, controlled by monitoring the RAS mutation load by liquid biopsy in RAS-mutated **MCRC** patients

A randomized phase II study with FOLFIRI-based 1st-line therapy with or without intermittent cetuximab

We, the undersigned, have read the Statistical Analysis Plan and agree that it contains all information required for statistical analysis of the data collected in the above-named noninterventional study.

| Autnor | Or. Christine Windemuth-Kleselbach (Statistics) |
|-------------------------|-------------------------------------------------|
| | DocuSigned by: |
| 16.09.2024 08:59 MESZ | a. Windemuk-Weselbal |
| Date | Signature |

**Sponsor** 

16.09.2024 | 12:46 MESZ Date

Hanno Härtlein DocuSigned by:

Signature

**National Coordinating Investigator** 

16.09.2024 | 14:28 MESZ Date

PD Dr. Alexander Baraniskin Prof. Dr. Alexander Baraniskin

Signature

-CEAD601C4E9D46E...

### **Table of contents**

| 1 | | of Abbreviationsduction | |
|---|---|---|---|
| _ | | Background | |
| 2 | | Study design | |
| 3 | | ysis data and patient populations | |
| | | Study objective | |
| | | Analysis populations | |
| | | Patient withdrawal(s) | |
| | 3.4 | Objectives | |
| 4 | | ods of analysis | |
| | | Hypotheses | |
| | | Statistical methods | |
| | | Statistical analysis | |
| | 4.3.1 | Baseline (anamnesis and one-time-only baseline examinations) | . 7 |
| | 4.3.2 | | |
| | 4.3.3 | Recurring examinations and lab assessments | ٤ . |
| | 4.3.4 | Study treatment | . ٤ |
| | 4.3.5 | Primary objective | ٤ . |
| | 4.3.6 | Secondary objectives (excluding safety) | . દ |
| | 4.3.7 | | |
| | 4.3.8 | End of study treatment, follow-up visits, and end of study | . 6 |
| | 4.3.9 | | |
| | 4.4 | Methods for handling missing data | 10 |
| | | Methods for handling inconsistent data | |
| | 4.6 | Methods for handling outliers | |
| | 4.7 | Methods for point and interval estimates | |
| | 4.8 | Validation of statistical methods | |
| | 4.9 | Methods for handling multicenter trial data | 10 |
| | 4.10 | Treatment interactions | |
| | 4.11 | Methods for handling repeated measurements | 10 |
| | 4.12 | Calculation of derived variables | 10 |
| | 4.13 | Use of baseline values | 11 |
| | 4.14 | Use of covariates | 11 |
| | 4.15 | Identification of fixed and random factors | 11 |
| | 4.16 | Subset analyses | 11 |
| | | Interim and follow-up analyses | |
| | | Study stopping rules | |
| | | Statistical significance levels | |
| | | Methods for handling dropouts and protocol violators | |
| | | Methods for handling more than two treatment groups | |
| | | Methods for handling concomitant medications | |
| | | Changes to the planned analyses | |
| 5 | Mocl | κ-ups for tables, listings, and figures | 13 |
| | 5.1 | Tables | |
| | 5.2 | Listings | |
| | | Figures | |
| 6 | | stical software | |
| 7 | | cal dictionaries | |
| 8 | | ng conventions | |
| 9 | | out format | |
| 10 | | of the tables, listings, and figures planned for the Final Statistical Report | |
| 11 | | pry table | |
| | | • | |

### 1 List of Abbreviations

| AE ALAT Alanine aminotransferase (also GPT for glutamate pyruvate transaminase) ASAT Aspartate aminotransferase (also GOT for glutamate oxaloacetate transaminase) BEAM(ing) Beads, emulsion, amplification, and magnetics (digital PCR) (β-)HCG (β-)HCG BRAF B-rapidly accelerated fibrosarcoma CA 19-9 CEA Carcinoembryonic antigen CR CR Complete response (m)CRC (metastatic) Colorectal cancer (e)CRF CRP C-reactive protein CT Computer tomography CTCAE Common Terminology Criteria of Adverse Events (version 5.0) ctDNA CTFG CInical Trail Facilitation Group ddPCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG EGFR Epidermal growth factor receptor EOT EOT EOT EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan F-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium International Statistical Classification of Diseases and Related Health Problems (10th revision from 2010) |
|---|
| transaminase) ASAT Aspartate aminotransferase (also GOT for glutamate oxaloacetate transaminase) BEAM(ing) Beads, emulsion, amplification, and magnetics (digital PCR) (β-)HCG (beta) Human chorionic gonadotropin BRAF B-rapidly accelerated fibrosarcoma CA 19-9 Carbohydrate antigen 19-9 CEA Carcinoembryonic antigen CR Complete response (m)CRC (metastatic) Colorectal cancer (e)CRF (electronic) Case report form CRP C-reactive protein CT Computer tomography CTCAE Common Terminology Criteria of Adverse Events (version 5.0) ctDNA Circulating cell-free tumor DNA CTFG Clinical Trail Facilitation Group ddPCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DpR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan F-FU Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| transaminase) ASAT Aspartate aminotransferase (also GOT for glutamate oxaloacetate transaminase) BEAM(ing) Beads, emulsion, amplification, and magnetics (digital PCR) (β-)HCG (beta) Human chorionic gonadotropin BRAF B-rapidly accelerated fibrosarcoma CA 19-9 Carbohydrate antigen 19-9 CEA Carcinoembryonic antigen CR Complete response (m)CRC (metastatic) Colorectal cancer (e)CRF (electronic) Case report form CRP C-reactive protein CT Computer tomography CTCAE Common Terminology Criteria of Adverse Events (version 5.0) ctDNA Circulating cell-free tumor DNA CTFG Clinical Trail Facilitation Group ddPCR Droplet Digital PCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DpR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan F-FU Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| oxaloacetate transaminase) BEAM(ing) (B-)HCG (beta) Human chorionic gonadotropin BRAF B-rapidly accelerated fibrosarcoma CA 19-9 CEA Carcinoembryonic antigen CR Complete response (m)CRC (metastatic) Colorectal cancer (e)CRF (electronic) Case report form CT CRP C-reactive protein CT COmputer tomography CTCAE Common Terminology Criteria of Adverse Events (version 5.0) ctDNA Circulating cell-free tumor DNA CTFG Clinical Trail Facilitation Group ddPCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DSMB Data and Safety Monitoring Board EC ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI Gamma-glutamyltransferase IC Inclusion Criterium International Statistical Classification of Diseases and Related |
| oxaloacetate transaminase) BEAM(ing) (β-)HCG (beta) Human chorionic gonadotropin BRAF B-rapidly accelerated fibrosarcoma CA 19-9 Carbohydrate antigen 19-9 CEA Carcinoembryonic antigen CR Complete response (m)CRC (metastatic) Colorectal cancer (e)CRF (electronic) Case report form CT CRP C-reactive protein CT Computer tomography CTCAE Circulating cell-free tumor DNA CTFG Clinical Trail Facilitation Group ddPCR Droplet Digital PCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DpR Depth of response DSMB Data and Safety Monitoring Board EC ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| BEAM(ing) (B-)HCG (beta) Human chorionic gonadotropin BRAF B-rapidly accelerated fibrosarcoma CA 19-9 Carbohydrate antigen 19-9 CEA Carcinoembryonic antigen CR Complete response (m)CRC (metastatic) Colorectal cancer (e)CRF (electronic) Case report form CRP C-reactive protein CT Computer tomography CTCAE Common Terminology Criteria of Adverse Events (version 5.0) ctDNA Circulating cell-free tumor DNA CTFG Clinical Trail Facilitation Group ddPCR Droplet Digital PCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan FFU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| (β-)HCG BRAF B-rapidly accelerated fibrosarcoma CA 19-9 CEA Carcinoembryonic antigen CR Complete response (m)CRC (e)CRF CP CT Computer tomography CTCAE Common Terminology Criteria of Adverse Events (version 5.0) CTCAE CIculating cell-free tumor DNA CTFG CInical Trail Facilitation Group ddPCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DSMB Data and Safety Monitoring Board EC EC Exclusion criterium ECG EGFR Epidermal growth factor receptor EOT EOT EOT EOT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| BRAF CA 19-9 Carbohydrate antigen 19-9 CEA Carcinoembryonic antigen CR Complete response (m)CRC (metastatic) Colorectal cancer (e)CRF (electronic) Case report form CRP C-reactive protein CT Computer tomography CTCAE Common Terminology Criteria of Adverse Events (version 5.0) ctDNA Circulating cell-free tumor DNA CTFG Clinical Trail Facilitation Group ddPCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DpR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR EDT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan F-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| CA 19-9 CEA Carcinoembryonic antigen CR Complete response (m)CRC (metastatic) Colorectal cancer (e)CRF (electronic) Case report form CRP C-reactive protein CT Computer tomography CTCAE Common Terminology Criteria of Adverse Events (version 5.0) ctDNA CIFC CICILIATI Facilitation Group ddPCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR EDT EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan ICD(10) International Statistical Classification of Diseases and Related |
| CEA Carcinoembryonic antigen CR Complete response (m)CRC (metastatic) Colorectal cancer (e)CRF (electronic) Case report form CRP C-reactive protein CT Computer tomography CTCAE Common Terminology Criteria of Adverse Events (version 5.0) ctDNA Circulating cell-free tumor DNA CTFG Clinical Trail Facilitation Group ddPCR Droplet Digital PCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DpR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| CR Complete response (m)CRC (metastatic) Colorectal cancer (e)CRF (electronic) Case report form CRP C-reactive protein CT Computer tomography CTCAE Common Terminology Criteria of Adverse Events (version 5.0) ctDNA Circulating cell-free tumor DNA CTFG Clinical Trail Facilitation Group ddPCR Droplet Digital PCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DpR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| (m)CRC (metastatic) Colorectal cancer (e)CRF (electronic) Case report form CRP C-reactive protein CT Computer tomography CTCAE Common Terminology Criteria of Adverse Events (version 5.0) ctDNA Circulating cell-free tumor DNA CTFG Clinical Trail Facilitation Group ddPCR Droplet Digital PCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DpR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| (e)CRF (electronic) Case report form CRP C-reactive protein CT Computer tomography CTCAE Common Terminology Criteria of Adverse Events (version 5.0) ctDNA Circulating cell-free tumor DNA CTFG Clinical Trail Facilitation Group ddPCR Droplet Digital PCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DPR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| CRP C-reactive protein CT Computer tomography CTCAE Common Terminology Criteria of Adverse Events (version 5.0) ctDNA Circulating cell-free tumor DNA CTFG Clinical Trail Facilitation Group ddPCR Droplet Digital PCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DpR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| CT Computer tomography CTCAE Common Terminology Criteria of Adverse Events (version 5.0) ctDNA Circulating cell-free tumor DNA CTFG Clinical Trail Facilitation Group ddPCR Droplet Digital PCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DpR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| CTCAE ctDNA Circulating cell-free tumor DNA CTFG Clinical Trail Facilitation Group ddPCR Droplet Digital PCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DpR Depth of response DSMB EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR EOT End of (study) treatment (m)FOLFIRI GGT Gamma-glutamyltransferase IC Inclusion Criterium Circulating cell-free tumor DNA Circulating cell-free tumor DNA Circulating cell-free tumor DNA Clinical Trail Facilitation Group Bound Adverse Events (version 5.0) Adverse Events (version 5.0) Circulating cell-free tumor DNA Clinical Trail Facilitation Group Board ECR Exclusion criterium Floor cacid Floor cacid, 5-FU, and irinotecan Fluorouracil Gamma-glutamyltransferase IC Inclusion Criterium International Statistical Classification of Diseases and Related |
| ctDNA Circulating cell-free tumor DNA CTFG Clinical Trail Facilitation Group ddPCR Droplet Digital PCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DpR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| CTFG Clinical Trail Facilitation Group ddPCR Droplet Digital PCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DpR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| ddPCR DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DpR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| DNA Deoxyribonucleic acid DPD Dihydropyrimidine dehydrogenase DpR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| DPD Dihydropyrimidine dehydrogenase DPR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| DpR Depth of response DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| DSMB Data and Safety Monitoring Board EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| EC Exclusion criterium ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| ECG Electrocardiogram ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| ECOG Eastern Cooperative Oncology Group EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| EGFR Epidermal growth factor receptor EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| EOT End of (study) treatment (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| (m)FOLFIRI (modified) Folinic acid, 5-FU, and irinotecan 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| 5-FU Fluorouracil GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| GGT Gamma-glutamyltransferase IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| IC Inclusion Criterium ICD(10) International Statistical Classification of Diseases and Related |
| ICD(10) International Statistical Classification of Diseases and Related |
| Health Problems (10" revision from 2010) |
| , |
| INR International normalized ratio |
| (m)ITT (modified) Intend-to-treat set |
| iv intravenous |
| KRAS Kirsten Rat Sarcoma Virus |
| LVEF Left ventricular ejection fraction |
| mAB Monoclonal antibodies |
| MedDRA Medical Dictionary for Regulatory Activities |
| NCI National Cancer Institute |
| NRAS Neuroblastoma RAS viral oncogene homolog |
| NYHA New York Heart Association |
| ORR Overall response rate |
| OS Overall survival |
| PCR Polymerase chain reaction |
| PD Progressive disease |
| PFS Progression free survival |
| PI3K Phosphatidylinositol-4,5-bisphosphate 3-kinase |
| PP Per-protocol |
| PR Partial response |
| PT Preferred terms |

| PTCA | Percutaneous transluminal coronary angioplasty |
|---------|------------------------------------------------------------------|
| (a)PTT | (activated) Partial thromboplastin time |
| RAS(wt) | Rat sarcoma (wild-type) |
| RECIST | Response Evaluation Criteria in Solid Tumors (version 1.1) |
| SAE | Serious adverse event |
| SD | Stable disease |
| SmPC | Summary of medicinal Product Characteristics |
| SOC | System organ class |
| SP | Safety population |
| TLF | Tables, listings, and figures |
| TFTS | Time to failure of treatment strategy |
| TNM | Tumor, node, and metastases (classification of malignant tumors) |
| UICC | Union for International Cancer Control |
| ULN | Upper limit of normal |
| VEGF | Vascular endothelial growth factor |
| WCRF | World Cancer Research Fund |
| WOCBP | Woman of childbearing potential |

#### 2 Introduction

#### 2.1 Background

Colorectal cancer (CRC) is the third most common cancer worldwide and its therapeutic management strongly depends on the disease stage and the genetic profile of the tumor. Due to improved diagnosis and introduction of new therapies including targeting therapies with anti-epidermal growth factor receptor (EGFR) or anti-vascular endothelial growth factor (VEGF) treatments, the CRC death rates declined over the past three decades.

Differentiating between right-sided and left-sided CRC, multiple randomized studies have consistently shown that primary tumor location in the right side is associated with minor response to anti-EGFR therapy despite Rat sarcoma wild-type (RASwt) status. Hence, the treatment with EGFR antibodies in first-line therapy is recommended for left-sided primary tumors with RASwt only.

Retrospective analyses of patients with RASwt metastatic CRC (mCRC) from the phase III trials CRYSTAL and FIRE-3 show that the administration of standard first-line chemotherapy with fluorouracil, folinic acid, and irinotecan (FOLFIRI) together with the monoclonal antibody (mAB) cetuximab had a markedly better prognosis on progression free survival (PFS), overall survival (OS), and overall response rate (ORR).

#### 2.2 Study design

This study is an open-label, prospective, randomized, and multicenter phase II trial that will evaluate the efficacy and safety of intermittent addition of cetuximab to a (modified) FOLFIRI-based first-line therapy to patients with RAS-mutant mCRC at diagnosis who convert to RASwt using monitoring of RAS mutation status by liquid biopsy. Maximum planned treatment duration amounts to 36 months with a total trial duration of 4.5 years.

#### 3 Analysis data and patient populations

In this section the planned statistical analyses will be outlined in accordance with the study protocol and with respect to the underlying data. The statistical methods will be described in detail and the Mock-ups of the tables, listings, and figures (TLF) to be used in the statistical report will be defined.

#### 3.1 Study objective

The aim of this randomized study is to evaluate whether patients with left-sides RAS-mutant mCRC at diagnosis will derive benefit from the adaption of adding cetuximab to the first-line therapy with FOLFIRI after RAS-mutation status has changed to wild-type and changing back

to FOLFIRI, as required, if RAS-mutation status has changed back to mutant, depending upon, and monitored by longitudinal ctDNA liquid biopsies.

### 3.2 Analysis populations

**Modified Intention to Treat (mITT)**: All randomized patients who received at least 1 dose, complete or incomplete, of study medication.

**Safety population (SP)** = mITT population.

**Per protocol (PP) population**: All randomized patients who received study treatment according to randomization and did not have major disqualifying protocol violations, i.e., did not violate any selection criterion.

#### 3.3 Patient withdrawal(s)

Patients will be encouraged to complete the study but may voluntarily withdraw from the study at any time. The investigator may also, with her/his discretion, withdraw the patient from participating in this study at any time, or the sponsor may discontinue the study. Reasons for early withdrawal from the study are documented in the electronic case report form (eCRF) as:

- Study closed/terminated,
- Patient is lost to follow-up,
- Patient died,
- Investigator's decision,
- Patient withdrew consent,
- Others such as medical advice or patient wish.

Patients withdrawn by withdrawal of informed consent, patient preference, or the investigator's decision, for reasons other than PD, will be defined as premature withdrawals.

#### 3.4 Objectives

### Primary objective:

 Evaluate efficacy in terms of PFS from the date of randomization in the study according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria in experimental and control arms.

#### Secondary objectives:

- OS in experimental and control arms from date of randomization,
- Time to failure of treatment strategy (TFTS) in experimental and control arms after randomization,
- PFS rate one year after date of randomization,
- Depth of response (DpR) in terms of reduction of tumor mass in experimental and control arms after of first-line treatment,
- Metastatic resections in experimental and control arms after first-line treatment,
- ORR defined as proportion of patients with partial response (PR) or complete response (CR) as best response in experimental and control arms after start of first-line treatment,
- Safety profile according to the National Cancer Institute's (NCI) Common Terminology Criteria of Adverse Events (CTCAE) version 5.0 criteria in experimental and control arms recorded from date of signature of informed consent.

#### Exploratory objectives (optional):

To identify driver mutations (e.g., BRAF, PI3k/AKT/mTOR etc.) in patients with PD under cetuximab therapy who remain RASwt in liquid biopsy,

 To compare the efficacy in terms of PFS in patients with conversion to RASwt in both BEAMing (standing for beads, emulsion, amplification, and magnetics) digital polymerase chain reaction (PCR) and Digital Droplet PCR (ddPCR) with those patients showing conversion to RASwt in ddPCR but not in BEAMing.

#### 4 Methods of analysis

### 4.1 Hypotheses

Initially, the hypothesis of this study was to show that the difference in PFS at twelve months between the experimental arm and control arm would amount to 20% meaning an increase from 30% to 50% (Hazard ratio = 0.5757). The estimated number of patients screened was 144 and the estimated number of randomized patients was 116.

#### 4.2 Statistical methods

Due to the actual small number of patients enlisted (seven) the study enrollment was closed. Most analyses will therefore be based on listings. Summary statistics of continuous variables like mean, standard deviation, and quantiles will not be provided. Derived variables like ORR, OS, and PFS will be shown as well and for time-to-event variables Kaplan-Meier plots will be given. A swimmer plot showing the treatment and response timeline for each patient will be added. Each listing will show the patient number, the arm into which the patient was randomized, and all relevant variables.

There will be no differentiation between the analysis populations.

### 4.3 Statistical analysis

In a first table we give an overview:

 General data such as number of patients, number of participating clinics, and analysis populations (Table 1).

### 4.3.1 Baseline (anamnesis and one-time-only baseline examinations)

All background data of the patients including demographics, relevant concomitant diseases and medication, and baseline characteristics from pre-screenings which are performed only once will be listed by patient number. Other baseline examinations and laboratory assessments will be summarized together with the same recurring examinations and assessments, respectively. The following listings are planned here:

- Inclusion criteria (Listing 1.1 to Listing 1.3),
- Exclusion criteria (Listing 2.1 to Listing 2.4),
- Eligibility for study participation as well as enrollment for screening phase and randomization (Listing 3),
- Patient characteristics like age, ethnic origin, and gender (Listing 4),
- Initial diagnosis of mCRC (Listing 5.1 to Listing 5.3),
- Relevant diseases according to the 10th revision of the International Statistical Classification of Diseases and Related Health Problems (ICD10) catalog (Listing 6),
- Relevant premedication (Listing 7.1) and concomitant medication (Listing 7.2),
- Baseline echocardiography with left ventricular ejection fraction (LVEF) (Listing 8),
- Tumor, nodes, and metastases classification of malignant tumors (TNM) staging at baseline (Listing 9),
- Baseline coagulation parameters international normalized ratio (INR) and partial thromboplastin time (PTT) (Listing 10),
- Baseline dihydropyrimidine dehydrogenase (DPD) deficiency (Listing 11)
- Baseline hepatitis serology (Listing 12).

#### 4.3.2 Randomization

All enrolled patients with conversion of mutant RAS as estimated centrally by liquid biopsy of cfDNA within the first 4 months (at week 4, 8, 12, or 16) and without PD as determined by CT scan will be randomized at week 8, for patients converting at week 4 or 8, and at week 16, for patients converting at week 12 or 16, directly after the CT scan in a 1:1 ratio to either experimental Arm A (switch arm) or control Arm B. Patients with PD before the randomization will not be considered for randomization.

The randomization into the respective treatment arm will be displayed together with the patient number in each listing.

### 4.3.3 Recurring examinations and lab assessments

Data gathered through examinations or assessments that are possibly not only performed at baseline such as electrocardiogram (ECG) as well as such that are planned in regular intervals including hematological and blood chemistry lab assessments, pregnancy tests, and tumor marker assessments are given here. An exception is the data obtained from RECIST assessments which belongs to the primary objective. The following listings will be included:

- Performed ECG assessments (Listing 13),
- Determined Eastern Cooperative Oncology Group (ECOG) performance statuses (Listing 14),
- Vital signs such as weight and heartrate (Listing 15),
- Hematological parameters hemoglobin, platelets, leukocytes, and neutrophils (Listing 16),
- Biochemical parameters including specific minerals, gamma-glutamyltransferase (GGT), aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), and C-reactive protein (CRP) (Listing 17.1 and Listing 17.2),
- Tumor marker parameters carcinoembryonic antigen (CEA) and carbohydrate antigen 19-9 (CA 19-9) (Listing 18).
- RAS mutation analyses performed on tumor tissue with possible detection of Kirsten Rat Sarcoma (KRAS) or neuroblastoma RAS viral oncogene homolog (NRAS) mutations (Listing 19),
- Taken blood samplings for liquid biopsy (Listing 20.1 and Listing 20.2),
- Beta human chorionic gonadotropin (β-HCG) pregnancy tests for women of childbearing potential (WOCBP) (Listing 21).

#### 4.3.4 Study treatment

All data concerning treatment cycles and administered chemotherapeutic treatments will be listed by patient number. The following listings are planned:

- General information such as start date, cycle number, and possible resections (Listing 22.1),
- Specific data on administration of irinotecan (Listing 22.2), folinic acid (Listing 22.3), fluorouracil (5-FU) (Listing 22.4 and Listing 22.5), and cetuximab (Listing 22.6).

These listings will be accompanied by:

 A swimmer plot visualizing the treatment (changes) together with points in time of response for each individual study participant (Figure 1).

#### 4.3.5 Primary objective

For the analysis concerning the primary objective the following three listings are given and considered for PFS:

• RECIST assessments (Listing 23.1) and observation of measurable and non-measurable (Listing 23.2) lesions via computer tomography (CT).

In addition.

• a listing containing PFS, OS, and TFTS (Listing 24)

will be created. Furthermore,

a Kaplan-Meier plot for PFS (Figure 2)

will be presented.

#### 4.3.6 Secondary objectives (excluding safety)

Due to the small number of patients neither all secondary objectives will be analyzed, nor full Kaplan-Meier methods will be applied to time-to-event analyses. Only OS,TFTS, and ORR will be considered. The first two named will be shown in the listing containing the primary objective PFS above, and in addition two Kaplan-Meier plots will be presented:

- a Kaplan-Meier plot for OS (Figure 3)
- a Kaplan-Meier plot for TFTS (Figure 4)

The remaining derived variable, ORR, will be given in

• a table displaying responses to study treatment together with ORR (Table 2).

#### 4.3.7 Exploratory objectives

Due to the small number of patients no explorative objective will be analyzed.

### 4.3.8 End of study treatment, follow-up visits, and end of study

Some data related to end of (study) treatment (EOT) or follow-ups such as AEs or lab assessments will already be listed in the corresponding listings. Remaining data will be included in the following listings:

- EOT with possible new tumor therapy (Listing 25),
- Follow-ups with changes to therapy (Listing 26.1) or performed surgeries (Listing 26.2),
- Date and reason for end of study (Listing 27).

#### **4.3.9 Safety**

Regarding the secondary objective safety, all adverse events (AEs) will be ordered by patient number and summarized in the following listings:

• Terminology and timeline of AE together with causality to study treatments as well as possible actions taken (Listing 28.1) and serious or special classification (Listing 28.2).

Optionally, if the number of AEs is sufficient, then the AEs will be analyzed in frequency tables including number of treatment-related AEs, number of AEs that cause permanent treatment discontinuation, system organ class (SOC) and preferred terms (PT) according to the Medical Dictionary for Regulatory Activities (MedDRA). The following tables will optionally be added:

 An AE overview (Table 4.1), number of AEs with respect to MedDRA grouping and NCI CTCAE grading (Table 4.2), and number of patients with AE by maximal grade with respect to MedDRA coding.

SAEs are classified as special if they involve pregnancy or medication error.

#### 4.4 Methods for handling missing data

Missing data will not be imputed.

#### 4.5 Methods for handling inconsistent data

Not applicable.

#### 4.6 Methods for handling outliers

Outliners will not be excluded from analysis.

### 4.7 Methods for point and interval estimates

Not applicable.

#### 4.8 Validation of statistical methods

Not applicable.

#### 4.9 Methods for handling multicenter trial data

Patients from all study centers will be pooled and tabulated as a single target group.

#### 4.10 Treatment interactions

There will be no analyses on treatment interactions, but interactions stated in the Summary of medicinal Product Characteristics (SmPC) of each study treatment are beside others:

- Folinic acid may increase the risk of toxicity associated with 5-FU which may be indicated by diarrhea or other gastrointestinal events; both must not be mixed for infusions.
- The combination of cetuximab and fluoropyrimidines such as 5-FU may increase risk of cardiac ischemia or hand-foot syndrome.
- There is no evidence that irinotecan and cetuximab influence each other. Further, the pharmacokinetic of irinotecan is not affected in combination with folinic acid and 5-FU.

#### 4.11 Methods for handling repeated measurements

No formal repeated measures analysis will be performed.

#### 4.12 Calculation of derived variables

First, we will clarify some notions regarding trial periods:

<u>Baseline/pre-screening phase</u> (within four weeks before start of treatment): First period of the trial where baseline examinations and baseline lab assessments are performed to confirm eligibility for study participation.

<u>Screening/pre-randomization phase</u> (begins with enrollment of patients and lasts for a maximum of sixteen weeks from start of standard first-line therapy with (m)FOLFIRI): Second period of the trial where conversion to RASwt is monitored and randomization is taking place if (early) conversions are confirmed.

Randomization/study treatment phase (begins with randomization and has a maximal duration of 36 months from start of first-line therapy): Third period where patients are treated with the respective study treatment according to their randomization into experimental Arm A or control Arm B.

Final assessment: Last assessment about four weeks after last treatment administration.

Follow-up: Time from last administration of study treatment until end of study

<u>Pre-cycle</u>: Notion for a treatment cycle in the pre-randomization phase.

Independent of the trail period, each (pre-)cycle has a duration of 14 days. The date of the eighth day of a cycle may be derived from given data as seventh day after the first day of that cycle.

<u>Pre-medication: All medication before first administration of any study treatment, i.e., before first pre-cycle.</u>

Primary and secondary derived variables are defined and calculated as follows:

<u>PFS</u>: Defined as being the time between date of randomization until date of progression according to RECIST v1.1 criteria or date of death from any cause, whichever occurs first. Any change in RAS mutation status without PD according to the RECIST criteria is not considered a PFS event. In patients without a PFS event, PFS will be censored on the last date they were known to be alive and progression-free (last valid tumor assessment) or at the start of a new anti-tumor therapy. Patients becoming eligible for surgery during study treatment will not be censored for PFS at this resection event.

OS: Defined as time from date of randomization until death from any cause. In patients without an OS event, OS will be censored on the last date they were known to be alive.

<u>ORR</u>: Defined as the proportion of randomized patients with CR or PR as best response since start of first-line therapy.

<u>TFTS</u>: Defined as the time from date of randomization to failure of treatment strategy, i.e., treatment discontinuation for any reason, including disease progression, withdrawal of consent, treatment toxicity, patient preference, loss to follow up, or death from any cause.

An AE will be called treatment-related if its occurrence is definitely, probably, or possibly related to the administration of any study treatment.

Note that a year is equal to 365 days, a month is equal to 30.4 days, and a week is equal to 7 days for duration calculations.

#### 4.13 Use of baseline values

The staging results of RECIST tumor assessments including date of assessment, size(s) of target tumor(s), or number of metastases at baseline are used for PFS analysis.

### 4.14 Use of covariates

Not applicable.

#### 4.15 Identification of fixed and random factors

Not applicable.

### 4.16 Subset analyses

No subgroup analyses are planned.

### 4.17 Interim and follow-up analyses

No interim analyses will be done due to the small number of participants. No follow-up analyses are planned.

### 4.18 Study stopping rules

The study may be discontinued at the discretion of the sponsor in any of the following events:

- Medical or ethnical reasons affecting the continued performance of the study (e.g., recommendations of the DSMB in the above-mentioned special stopping rules after randomization of the first twenty patients and screening of the first fifty patients, respectively),
- Difficulties in the recruitment of patients,
- Inefficacy of the study treatment,
- Occurrence of AEs previously unknown in respect of their nature, severity, and duration or unexpected incidence of known AEs.

### 4.19 Statistical significance levels

Not applicable.

#### 4.20 Methods for handling dropouts and protocol violators

Patients withdrawn from the study for reasons stated in section 3.3 will not be replaced.

For patients considered to be significantly noncompliant by the investigator or sponsor with the requirements of the protocol, i.e., protocol violations such as pregnancy, the treatment will be permanently discontinued. Other reasons for permanent treatment discontinuation for a patient include withdrawal criteria and:

- Three years of study treatment,
- Patient experiences PD,
- Patient experiences unacceptable toxicity or an adverse experience that would, in the investigator's or sponsor's judgment, make continued administration of the study regimen an unacceptable risk,
- Situations requiring a therapeutic intervention not permitted by the treatment plan,
- Development of an intercurrent illness or situation which would, in the judgement of the investigator, affect assessments of clinical status and study endpoints to a significant degree,
- Specific request of the sponsor.

Patients for whom the treatment is permanently discontinued will remain in the study unless withdrawal. All patients with permanent treatment discontinuation, except for withdrawal of informed consent, lost to follow-up, or death, will be followed up as planned.

#### 4.21 Methods for handling more than two treatment groups

Not applicable.

### 4.22 Methods for handling concomitant medications

Concomitant medications will be listed in Listing 6.2. There will be no analysis of their impact on study treatment or outcome.

### 4.23 Changes to the planned analyses

Due to the small number of patients, most analyses are shown in listings. Not all study objectives can be considered.

### 5 Mock-ups for tables, listings, and figures

The following TLF are planned. The fields marked in checked grey (listings) and the grey text in curly braces (tables) show the programmer where the parameter to be analyzed may be found and will not appear in the report.

Regarding listings, alternative choices such as yes or no, male or female, and positive or negative will not be displayed, but units will be given as shown below. Furthermore, abbreviations listed in chapter 1 will be used for legibility.

#### **5.1** Tables

Table 1: General data

| Populations | [N, %] |
|--------------------------------------------|-------------|
| Number of patients | xx (100.00) |
| Number of patients in analysis populations | |
| mITT=SP | |
| PP | |
| Number of patients in treatment arms | |
| A | |
| В | |
| Number of participating clinics | |

### Table 2: Patients' first conversion to RAS wild-type

| | Time fro | ime from baseline sampling until first detection of RASwt [days] | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | N | Mean | STD | Min | Q1 | Median | Q3 | Max | NMiss |
| Α | | | | | | | | | |
| В | | | | | | | | | |
| Total | | | | | | | | | |

# Table 3: Responses

| Responses according to RECIST v1.1 criteria including Overall response rate (ORR) | Arm A [N, %] | Arm B [N, %] | Total [N, %] |
|---|---|---|---|
| Number of randomized patients | | | |
| Most recent response | | | |
| Complete response (CR) | | | |
| Partial response (PR) | | | |
| Stable disease (SD) | | | |
| Progressive disease (PD) | | | |
| Best response | | | |
| Complete response (CR) | | | |
| Partial response (PR) | | | |
| Stable disease (SD) | | | |
| Progressive disease (PD) | | | |
| Overall response | | | |
| CR or PR (ORR) | | | |

### (Optionally) Table 4.1: AEs - overview

| Overview | 5-FU [N, %] | Folinic acid<br>[N,%] | Irinotecan<br>[N,%] | Cetuximab<br>[N, %] | Total [N, %] |
|---|---|---|---|---|---|
| Number of patients in mITT | | | | | |
| Patients with any AE | | | | | |
| Patients with AEs by maximal grade | | | | | |
| Grade 1 | | | | | |
| Grade 2 | | | | | |
| Grade 3 | | | | | |
| Grade 4 | | | | | |

| Protocol | Codo | NΙα | 1212000 | ١ |
|----------|------|------|---------|---|
| Protocor | Code | INO. | 4213000 | , |

MoLiMoR

EudraCT-No. 2019-003714-14

| One de E |
|--------------------------------------------------|
| Grade 5 |
| Number of AEs |
| Patients with treatment-related AEs |
| Number of treatment-related AEs |
| Patients with any SAE |
| Patients with SAEs by seriousness criteria |
| Death |
| Life-threatening |
| Hospitalization |
| Persistent or significant disability/incapacity |
| Congenital anomaly/birth defect |
| Important medical event |
| Number of SAEs |
| Patients with any special AE |
| Patients with special AEs by speciality criteria |
| Pregnancy |
| Medication error |
| Number of special AEs |
| Patients with AEs leading to discontinuation |
| Number of AEs leading to discontinuation |

### (Optionally) Table 4.2: AEs - System Organ Class (SOC) and Preferred Term (PT) by NCI CTCAE grade

| | | NCI C | TCAE | Total | | | | |
|---------------|----|-------|------|-------|---|---|---|-----|
| SOC | PT | 1 | 2 | 3 | 4 | 5 | N | % |
| Number of AEs | | | | | | | | 100 |

| SOC1 | |
|------|------|
| | PT11 |
| | PT12 |
| SOC2 | |
| | PT21 |
| | PT22 |

### (Optionally) Table 4.3: AEs - number of patients with respect to System Organ Class (SOC) and Preferred Term (PT) by maximal NCI CTCAE grade

| | | Maxin | nal NCI | CTCA | E grad | е | Total | |
|---|---|---|---|---|---|---|---|---|
| SOC | PT | 1 | 2 | 3 | 4 | 5 | N | % |
| Number of patients with any AE | | | | | | | | 100 |
| SOC1 | | | | | | | | |
| | PT11 | | | | | | | |
| | PT12 | | | | | | | |
| SOC2 | | | | | | | | |
| | PT21 | | | | | | | |
| | PT22 | | | | | | | |

# 5.2 Listings

# Eligibility criteria:

### Listing 1.1: Inclusion criteria - legend

| Abbreviation | Full text |
|---|---|
| IC 01 | Histologically confirmed, UICC stage IV adenocarcinoma of the left-sided colon or rectum with metastases, primarily non-resectable, confirmed RAS mutations proven in the primary tumor or metastasis (KRAS and NRAS exon 2, 3, 4) |
| IC 02 | Age ≥ 18 years on day of signing informed consent |
| IC 03 | No previous chemotherapy for metastatic disease (1-2 cycles FOLFIRI or mFOLFIRI are permitted before enrollment until RAS status is determined) |
| IC 04 | Patient is suitable for chemotherapy administration |
| IC 05 | ECOG performance status 0-1 |
| IC 06 | Consent to liquid biopsy and mutation analysis |
| IC 07 | Estimated life expectancy > 3 months |
| IC 08 | Presence of at least one measurable reference lesion according to the RECIST v 1.1 criteria (chest CT and abdominal CT four weeks or less before enrollment) |
| IC 09 | Adequate bone marrow function defined as: Leukocytes 3.0 x 109/L with neutrophils 1.5 x 109/L, thrombocytes 100 x 109/L, and hemoglobin 9 g/dL |
| IC 10 | Adequate hepatic function defined as: Serum bilirubin 1.5 x ULN, ALAT, and ASAT 2.5 x ULN (in the presence of hepatic metastases, ALAT and ASAT 5 x ULN) |
| IC 11 | Adequate renal function defined as: Creatinine clearance ≥ 50 mL/min |
| IC 12 | Adequate cardiac function defined as: Normal ECG and echocardiogram with a LVEF of 55% |
| IC 13 | INR < 1.5 and activated PTT (aPTT) < 1.5 x ULN (patients without anticoagulation). Therapeutic anticoagulation is allowed if INR and aPTT have remained stable within the therapeutic range for at least two weeks |
| IC 14 | Time interval of at least six months since last administration of any previous neoadjuvant/adjuvant chemotherapy or radio chemotherapy of the primary tumor in curative treatment intention to start of first-line treatment |
| IC 15 | Any relevant toxicities of prior treatments must have resolved to grade ≤ 1 according to the CTCAE (version 5), except alopecia |
| IC 16 | WOCBP should have a negative urine pregnancy test within 72 hours prior to receiving the first dose of study medication |
| IC 17 | Highly effective contraception for both male and female patients throughout the study and for at least three months after last dose of study medication administration if the risk of conception exists. Highly effective contraception must be in line with the definition of the CTFG recommendation |
| IC 18 | Signed written informed consent and capacity to understand the informed consent |
| IC 19 | Date of signing written informed consent |

# Listing 1.2: Inclusion criteria 01-09

| patient.pa retient_no | registration.registration | patient.pati | patient.pati | patient.pati | patient.pati | patient.pati | patient.pati | patient.pati | patient.pati | patient.pati |
|---|---|---|---|---|---|---|---|---|---|---|
| | _arm_randomized | ent_ic_01 | ent_ic_02 | ent_ic_03 | ent_ic_04 | ent_ic_05 | ent_ic_06 | ent_ic_07 | ent_ic_08 | ent_ic_09 |
| Patient | Arm | IC 01 | IC 02 | IC 03 | IC 04 | IC 05 | IC 06 | IC 07 | IC 08 | IC 09 |
| No. | | [yes/no] | [yes/no] | [yes/no] | [yes/no] | [yes/no] | [yes/no] | [yes/no] | [yes/no] | [yes/no] |

# Listing 1.3: Inclusion criteria 10-19

| patient.p<br>atient_no | registration.registrati<br>on_arm_randomized | | | | | | | | | | patient.patie<br>nt_ic_ic_date |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient<br>No. | Arm | IC 10<br>[yes/no] | IC 11<br>[yes/no] | IC 12<br>[yes/no] | IC 13<br>[yes/no] | IC 14<br>[yes/no] | IC 15<br>[yes/no] | IC 16<br>[yes/no/na<br>] | IC 17<br>[yes/no/na<br>] | IC 18<br>[yes/no] | IC 19<br>[DDMMMYY] |

# Listing 2.1: Exclusion criteria - legend

| Abbreviation | Full text |
|---|---|
| EC 01 | Right-sided mCRC |
| EC 02 | Primarily resectable metastases |
| EC 03 | Previous chemotherapy for the colorectal cancer except for adjuvant treatment, completed at least six months before entering the study (1-2 cycles FOLFIRI or mFOLFIRI are permitted before enrollment) |
| EC 04 | Patients with known brain metastases |
| EC 05 | Symptomatic peritoneal carcinosis |
| EC 06 | Progressive disease before randomization |
| EC 07 | History of acute or subacute intestinal occlusion, inflammatory bowel disease, immune colitis, or chronic diarrhea |
| EC 08 | Grade II heart failure (NYHA classification), Myocardial infarction, balloon angioplasty (PTCA) with or without stenting, and cerebral vascular accident/stroke within the past twelve months before enrollment, unstable angina pectoris, serious cardiac arrhythmia according to investigator's judgment requiring medication |
| EC 09 | Medical or psychological impairments associated with restricted ability to give consent or not allowing conduct of study |
| EC 10 | Active infection with hepatitis B or C |
| EC 11 | Additional cancer; exceptions include adequately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy without evidence of recurrence |
| EC 12 | Uncontrolled hypertension |
| EC 13 | Marked proteinuria (nephrotic syndrome) |
| EC 14 | Arterial thromboembolism or severe hemorrhage within six months prior to randomization (with exception of tumor bleeding before tumor resection surgery) |
| EC 15 | Hemorrhagic diathesis or tendency towards thrombosis |
| EC 16 | Participation in a clinical study or experimental drug treatment within thirty days prior to study |
| EC 17 | Known hypersensitivity or allergic reaction to any of the study medications |
| EC 18 | Severe, non-healing wounds, ulcers, bone fractures, or an infection requiring systematic therapy |
| EC 19 | Known history of alcohol or drug abuse |
| EC 20 | Known complete DPD deficiency (phenotype and/or genotype test) (patients with partial DPD deficiency may be included in this clinical trial at the discretion of the investigator and should receive a reduced starting 5-FU dose); known glucuronidation deficiency (Gilbert's syndrome) (specific screening not required) |
| EC 21 | Absent or restricted legal capacity |
| EC 22 | For female patients only: Pregnancy (absence to be confirmed by ß-HCG test) or lactating |

### Listing 2.2: Exclusion criteria 01-08

| patient.pati<br>ent_no | registration.registration_a<br>rm_randomized | patient.patie<br>nt_ec_01 | patient.patie<br>nt_ec_02 | patient.patie<br>nt_ec_03 | patient.patie<br>nt_ec_04 | patient.patie<br>nt_ec_05 | patient.patie<br>nt_ec_06 | patient.patie<br>nt_ec_07 | patient.patie<br>nt_ec_08 |
|---|---|---|---|---|---|---|---|---|---|
| Patient No. | Arm | EC 01<br>[yes/no] | EC 02<br>[yes/no] | EC 03<br>[yes/no] | EC 04<br>[yes/no] | EC 05<br>[yes/no] | EC 06<br>[yes/no] | EC 07<br>[yes/no] | EC 08<br>[yes/no] |

# Listing 2.3: Exclusion criteria 09-15

| patient.patie<br>nt_no | registration.registration_arm<br>_randomized | patient.patient<br>_ec_09 | patient.patient<br>_ec_10 | patient.patient<br>_ec_11 | patient.patient<br>_ec_12 | patient.patient<br>_ec_13 | patient.patient<br>_ec_14 | patient.patient<br>_ec_15 |
|---|---|---|---|---|---|---|---|---|
| Patient No. | Arm | EC 09 [yes/no] | EC 10 [yes/no] | EC 11 [yes/no] | EC 12 [yes/no] | EC 13 [yes/no] | EC 14 [yes/no] | EC 15 [yes/no] |

### Listing 2.4: Exclusion criteria 16-22

| patient.patie<br>nt_no | registration.registration_arm<br>_randomized | patient.patient<br>_ec_16 | patient.patient<br>_ec_17 | patient.patient<br>_ec_18 | patient.patient<br>_ec_19 | patient.patient<br>_ec_20 | _ec_21 | patient.patient<br>_ec_22 |
|---|---|---|---|---|---|---|---|---|
| Patient No. | Arm | EC 16 [yes/no] | EC 17 [yes/no] | EC 18 [yes/no] | EC 19 [yes/no] | EC 20 [yes/no] | EC 21 [yes/no] | EC 22<br>[yes/no/na] |

### Listing 3: Eligibility, enrollment, and randomization

| patient.patie<br>nt_no | patient.patient_study_eligibility | enrollment.enrollment_enrollment_date | registration.registration_regi<br>stered_at | registration.registration_arm_randomi<br>zed |
|---|---|---|---|---|
| Patient No. | Eligible for participation [yes/no] | Date of enrollment for screening phase | Date of randomization | Randomized into study arm |

# Patient characteristics and initial diagnosis:

# **Listing 4: Patient demographics**

| | registration.registration_arm_randomized | | baseline.baseli<br>ne_bodysize, | baseline.baseli<br>ne_bodyweight | | patient.patient_<br>wocbp | anamnesis.ana<br>mnesis_ethnic | patient.patient_protocol_v<br>ersion |
|---|---|---|---|---|---|---|---|---|
| Patient<br>No. | Arm | Age<br>[years] | Height [cm] | Weight [kg] | Sex<br>[female/male] | WOCBP<br>[yes/no] | Ethnic origin | Protocol version at informed consent [version] |

# Listing 5.1: Initial diagnosis of mCRC - TNM staging

| | registration.registrat<br>ion_arm_randomize<br>d | | anamnesis.anamn<br>esis_tnm_perform<br>ed | | | | | anamnesis.<br>anamnesis_<br>tnm_stage |
|---|---|---|---|---|---|---|---|---|
| Patient<br>No. | Arm | Date of initial<br>diagnosis | TNM staging performed at initial diagnosis [yes/no] | anamnesis.anamn<br>esis_tnm_t_prefix<br>Prefix | Classific anamnesis.ana mnesis_tnm_t T | anamnesis.ana | anamnesis.ana<br>mnesis_tnm_m<br>M | Stage |

# Listing 5.2: Initial diagnosis of mCRC - resection

| patient.patie<br>nt_no | registration.registratio<br>n_arm_randomized | anamnesis.anamnesis_resection_done | anamnesis.anamnesis_resectio<br>n_date(_nd) | anamnesis.anamnesis_resecti<br>on_status(_nd) |
|---|---|---|---|---|
| Patient No. | Arm | Primary tumor resected before study inclusion [yes/no] | Date of resection | Resection status |

# Listing 5.3: Initial diagnosis of mCRC - RAS mutation analysis

| patient.<br>patient<br>_no | registratio<br>n.registrati<br>on_arm_ra<br>ndomized | anamnesis.anamnesis_ras<br>_mutation_performed | anamnesis.anamnesis_ra s_mutation_m(_spec), anamnesis.anamnesis_ra s_mutation_m_n(_spec) | anamnesis.an<br>amnesis_ras_<br>mutation_stat<br>us | anamnesis.<br>anamnesis<br>_kras | anamnesis.anamn<br>esis_kras_mutatio<br>n_list | | anamnesis.anamn<br>esis_nras_mutatio<br>n_list |
|---|---|---|---|---|---|---|---|---|
| Patient<br>No. | Arm | RAS mutation analysis performed on tumor tissue [yes/no] | RAS mutation analysis<br>method | RAS mutation<br>status<br>[wt/mutant] | KRAS<br>detected<br>[yes/no] | Exon(s) and<br>Codon(s) of<br>KRAS mutation(s) | NRAS<br>detected<br>[yes/no] | Exon(s) and<br>Codon(s) of<br>NRAS mutation(s) |

# Medical history and relevant medications:

### **Listing 6: Medical history**

| patient.patie<br>nt_no | registration.registration_arm_r<br>andomized | anamnesis.anamnesis_con<br>_diseases | icd10_en2010_code.de<br>scription | disease.disease<br>_start | disease.diseas<br>e_end | disease.disease_end_<br>ongoing |
|---|---|---|---|---|---|---|
| Patient No. | Arm | Relevant concomitant diseases [yes/no] | Disease according to ICD10 | Start date | Stop date | Ongoing [yes/no] |

### Listing 7.1: Relevant medication - premedication

| patien<br>t.patie<br>nt_no | registratio<br>n.registrati<br>on_arm_ra<br>ndomized | anamnesis<br>.anamnesi<br>s_prev_m<br>edications | tion.me | tion.me | medication<br>.medicatio<br>n_indicatio<br>n(_spec) | | | | | medicati<br>on.medic<br>ation_fre<br>quency | medica<br>tion.me<br>dication<br>_route | tion.me |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patie<br>nt No. | Arm | Relevant<br>premedica<br>tion<br>[yes/no] | Preme<br>dication<br>treatme<br>nt | Start<br>date | Indication | medication<br>.medicatio<br>n_dose<br>Quantity | medication.me<br>dication_dose_<br>unit<br>Unit | Dose medication.me dication_dose_ na Unknown | medication.medic<br>ation_dose_requi<br>red<br>As required | Frequen<br>cy | Route | Stop<br>date |

# Listing 7.2: Relevant medication - concomitant medication

| | registrati<br>on.regist<br>ration_ar<br>m_rando<br>mized | precycle.prec<br>ycle_no,<br>therapycycle.t<br>herapycycle_<br>no | precycle.precycle_prev<br>_medications,<br>therapycycle.therapycy<br>cle_prev_medications | medic<br>ation.<br>medic<br>ation_<br>drug | medic<br>ation.<br>medic<br>ation_<br>start | medicati<br>on.medic<br>ation_ind<br>ication(_<br>spec) | | | | | medica<br>tion.me<br>dication<br>_freque<br>ncy | medic<br>ation.<br>medic<br>ation_<br>route | medica<br>tion.me<br>dicatio<br>n_stop |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patie<br>nt<br>No. | Arm | Point in time | Concomitant<br>medication changes<br>since last study<br>treatment [yes/no] | Medic<br>ation<br>treat<br>ment | Start<br>date | Indicatio<br>n | medicati<br>on.medic<br>ation_do<br>se<br>Quantity | medication .medicatio n_dose_u nit Unit | medicati on.medic ation_do se_na Unknown | medication. medication_ dose_requir ed As required | Freque<br>ncy | Route | Stop<br>date |
| | | Pre-cycle 1 | | | | | | | | | | | |
| | | Cycle 1 | | | | | | | | | | | |

### Baseline only examinations:

# Listing 8: Baseline echocardiography

| patient.pati<br>ent_no | registration.registration_<br>arm_randomized | baseline.baseline_ec<br>hocardio_done | baseline.baseline_echoca<br>rdio_nd(_spedc) | baseline.baseline_ec<br>hocardio_date | baseline.baseline_ec<br>hocardio_lvef | baseline.baseline_ech<br>ocardio_result |
|---|---|---|---|---|---|---|
| Patient<br>No. | Arm | Echocardiography performed [yes/no] | Reason if no | Date of echocardiography | LVEF [%] | Clinical significance |
| 1 | | | i e | | | |

### Listing 9: Baseline TNM staging

| patient.pa<br>tient_no | registration.registration<br>_arm_randomized | baseline.baselin<br>e_tnm_done | baseline.baseline_t<br>nm_nd(_spec) | baseline.baseli<br>ne_tnm_date | | | | |
|---|---|---|---|---|---|---|---|---|
| Patient<br>No. | Arm | TNM staging<br>performed<br>[yes/no] | Reason if no | Date of TNM<br>staging | baseline.baseline<br>tnm_t_prefix<br>Prefix | Classifice baseline.base line_tnm_t T | baseline.base line_tnm_n N | baseline.basel<br>ine_tnm_m<br>M |
| | | | _ | _ | | | | |

### Baseline only laboratory assessments:

### Listing 10: Baseline coagulation parameters

| patient.pati<br>ent_no | registration.registration_ar<br>m_randomized | lab_val_co.lab_val_c<br>o_lab_done | lab_val_co.lab_val_c<br>o_reason(_spec) | lab_val_co.lab_val_co<br>_date | lab_val_co.lab_val_c<br>o_inr_value | lab_val_co.lab_val_c<br>o_ptt_value |
|---|---|---|---|---|---|---|
| Patient No. | Arm | Coagulation done<br>[yes/no] | Reason if no | Date of coagulation sampling | INR | PTT [s] |

### **Listing 11: Baseline DPD deficiency**

| patient.patient<br>_no | registration.registration_arm<br>_randomized | baselab.baselab_dpd_done | baselab.baselab_dpd_reason(<br>_spec) | baselab.baselab_dpd_<br>date | baselab.baselab_dpd_r<br>esult |
|---|---|---|---|---|---|
| Patient No. | Arm | Test for DPD deficiency performed [yes/no] | Reason if no | Date for DPD deficiency test | Test result |

# Listing 12: Baseline hepatitis serology

| patient.pati<br>ent_no | registration.registration_ar<br>m_randomized | baselab.baselab_sero<br>logical_done | baselab.baselab_serologi<br>cal_nd(_spedc) | baselab.baselab_ser<br>ological_date | baselab.baselab_ser<br>ological_hbv | baselab.baselab_ser<br>ological_hcv |
|---|---|---|---|---|---|---|
| Patient No. | Arm | Serological tests performed [yes/no] | Reason if no | Date of serological tests | Hepatitis B<br>[positive/negative] | Hepatitis C [positive/negative] |

### Electrocardiogram assessments:

# Listing 13: ECG assessments

| patient.patie<br>nt_no | registra<br>tion.reg<br>istratio<br>n_arm_<br>random<br>ized | precycle.pr<br>ecycle_no,<br>therapycyc<br>le.therapyc<br>ycle_no | precycle.precycle_ecg_<br>performed. | baseline.baseline_ecg_nd(_spedc), precycle.precycle_ecg_nd(_spedc), therapycycle.therapycycle_ecg_nd(_ | precycle.precycle_ecg_date, | baseline.baseline_ecg_result, precycle.precycle_ecg_result, therapycycle.therapycycle_ec g_result |
|---|---|---|---|---|---|---|
| Patient No. | Arm | Point in time | ECG performed [yes/no] | Reason if no | Date of ECG | Clinical significance |
| | | Baseline | | | | |
| | | Pre-cycle | | | | |
| | | 1 | | | | |
| | | ••• | | | | |
| | | Cycle 1 | | | | |

### Eastern Cooperative Oncology Group performance statuses:

# **Listing 14: ECOG performance statuses**

| patient.patie<br>nt_no | registration.regi<br>stration_arm_ra<br>ndomized | precycle.precycle_no, therapycycle.therapycycle_cycle_n o | baseline.baseline_ecog_date, precycle.precycle_ecog_date(_nd), therapycycle.therapycycle_w1_ecog_date(_nd), therapycycle.therapycycle_w2_ecog_date(_nd), eot.eot_date, followup.followup_date | baseline.baseline_ecog, precycle.precycle_ecog, therapycycle.therapycycle_w1_ecog, therapycycle.therapycycle_w2_ecog, eot.eot_ecog, followup.followup_ecog |
|---|---|---|---|---|
| Patient No. | Arm | Point of time | Date of ECOG evaluation | ECOG performance status |
| | | Baseline | | |
| | | Pre-cycle 1 | | |
| | | Cycle 1 | | |
| | | EOT | | |
| | | Follow-up 1 | | |

# Vital signs examinations:

# **Listing 15: Vital signs**

| patie<br>nt.pat<br>ient_<br>no | registr<br>ation.r<br>egistr<br>ation_r<br>arm_r<br>ando<br>mized | precycle.<br>precycle<br>_no,<br>therapyc<br>ycle.ther<br>apycycle<br>_no | baseline.b aseline_vit al, precycle.pr ecycle_vit al, therapycyc le.therapyc ycle_w1_vi tal, therapycyc le.therapycyc le.therapyc ycle_w2_vi tal | baseline.baseline _vital_nd(_spec), precycle.precycle _vital_nd(_spec), therapycycle_ex am_performed, therapycycle.ther apycycle_w1_vit al_nd(_spec), therapycycle.ther apycycle_w2_vit al_nd(_spec) | baseline.baseline_v | baseline.base line_bodywei ght, precycle.prec ycle_bodywei ght, therapycycle.t herapycycle_ w1_bodyweig ht, therapycycle.t herapycycle.t herapycycle.t herapycycle.t herapycycle.t herapycycle.t herapycycle.t herapycycle.t | baseline.base line_body_te mp, precycle.prec ycle_body_te mp, therapycycle.t herapycycle_ w1_body_tem p, therapycycle.t herapycycle.t herapycycle.t herapycycle.t p, | baseline.baseli ne_bloodpress ure_s, precycle.precyc le_bloodpressu re_s, therapycycle.th erapycycle_w1 _bloodpressure _s, therapycycle.th erapycycle.th erapycycle.th erapycycle.th erapycycle.sy2 _bloodpressure _s | baseline.baseli ne_bloodpress ure_d, precycle.precyc le_bloodpressu re_d, therapycycle.th erapycycle_w1 _bloodpressure _d, therapycycle.th erapycycle.th erapycycle.th erapycycle.th erapycycle.d | baseline.ba<br>seline_puls<br>e,<br>precycle.pre<br>cycle_pulse<br>,<br>therapycycl<br>e.therapycy<br>cle_w1_pul<br>se,<br>therapycycl<br>e.therapycycl<br>e.therapycycl<br>e.therapycycl<br>se |
|---|---|---|---|---|---|---|---|---|---|---|
| Patie<br>nt<br>No. | Arm | Point in time | Vital signs<br>examined<br>[yes/no] | Reason if no | Date of examination | Weight [kg] | Temperature<br>[°C] | Blood pressure<br>(systolic)<br>[mmHg] | Blood pressure<br>(diastolic)<br>[mmHg] | Heartrate<br>[per min] |
| | | Baseline | | | | | | | | |
| | | Pre-cycle<br>1 | | | | | | | | |
| | | Cycle 1 | | | | | | | | |

### Hematological and blood chemistry laboratory assessments:

### Listing 16: Hematological lab assessments

| patient. patient _no | registration.regis<br>tration_arm_ran<br>domized | precycle.pre<br>cycle_no,<br>therapycycl<br>e.therapycy<br>cle_no | | lab_val_he.lab_<br>val_he_reason(<br>_spec) | lab_val_he.<br>lab_val_he<br>_date | lab_val_he.lab_v<br>al_he_haemoglob<br>in_value | lab_val_he.lab<br>_val_he_platel<br>_et_value | | lab_val_he.lab_v<br>al_he_neutrophil<br>t_value |
|---|---|---|---|---|---|---|---|---|---|
| Patient<br>No. | Arm | Point in time | Laboratory<br>hematology<br>done [yes/no] | Reason if no | Date of hematology sampling | Hemoglobin<br>[g/dL] | Platelets<br>[10 <sup>9</sup> /L] | Leukocytes<br>[10 <sup>9</sup> /L] | Neutrophils<br>(total) [10 <sup>9</sup> /L] |
| | | Baseline | | | | | | | |
| | | Pre-cycle 1 | | | | | | | |
| | | Cycle 1 | | | | | | | |
| | | EOT | | | | | <u>-</u> | | |

### Listing 17.1: Blood chemistry lab assessments - first part

| patien<br>t.patie<br>nt_no | registratio<br>n.registrati<br>on_arm_ra<br>ndomized | precycle.precyc<br>le_no,<br>therapycycle.th<br>erapycycle_no | lab_val_cc.lab_v<br>al_cc_lab_done | lab_val_c<br>c.lab_val<br>_cc_reas<br>on(_spec) | lab_val_c<br>c.lab_val_<br>cc_date | lab_val_cc.la<br>b_val_cc_sod<br>ium_value | lab_val_cc.lab<br>_val_cc_potas<br>_sium_value | lab_val_cc.lab_<br>val_cc_magnes<br>ium_value | lab_val_cc.lab<br>_val_cc_calci<br>_um_value | lab_val_cc.l<br>ab_val_cc_<br>got_value |
|---|---|---|---|---|---|---|---|---|---|---|
| Patie nt No. | Arm | Point in time | Laboratory blood chemistry done [yes/no] | Reason if no | Date of chemistry sampling | Sodium<br>[mval/L] | Potassium<br>[mmol/L] | Magnesium<br>[mmol/L] | Calcium<br>[mmol/L] | ASAT [U/L] |
| | | Baseline | | | | | | | | |
| | | Pre-cycle 1 | | | | | | | | |
| | | Cycle 1 | | | | | | | | |
| | | EOT | · | | | | | | | |

# Listing 17.2: Blood chemistry lab assessments - second part

| patien<br>t.patie<br>nt_no | registratio<br>n.registrati<br>on_arm_ra<br>ndomized | lab_val_cc<br>.lab_val_c<br>c_date | lab_val_cc.l<br>ab_val_cc_<br>gpt_value | lab_val_cc.lab_v<br>al_cc_alkphosph<br>atase_value | lab_val_cc.la<br>b_val_cc_bili<br>rubint_value | | lab_val_cc.la<br>b_val_cc_ure<br>a_value | lab_val_cc.lab_<br>val_cc_creatini<br>ne_value | lab_val_cc.lab_<br>val_cc_creatini<br>nec_value | lab_val_cc.la<br>b_val_cc_cr<br>p_value |
|---|---|---|---|---|---|---|---|---|---|---|
| Patie<br>nt No. | Arm | Date of<br>chemistry<br>sampling | ALAT [U/L] | Alkaline<br>phosphatase<br>[U/L] | Bilirubin<br>(total) | GGT [U/L] | Urea [mg/dL] | Creatinine<br>[mg/dL] | Creatinine-<br>clearance<br>[mL/s] | CRP [mg/dL] |

### Tumor tissue analyses:

### **Listing 18: Tumor markers lab assessments**

| patient.pa<br>tient_no | registration.registr<br>ation_arm_rando<br>mized | precycle.precycle_no,<br>therapycycle.therapyc<br>ycle_no | lab_val_tm.lab_val<br>_tm_lab_done | lab_val_tm.lab_val_t<br>m_reason(_spec) | lab_val_tm.lab_<br>val_tm_date | lab_val_tm.lab_val<br>_tm_cea_value | lab_val_tm.lab_val_t<br>m_ca199_value |
|---|---|---|---|---|---|---|---|
| Patient<br>No. | Arm | Point in time | Laboratory tumor<br>markers done<br>[yes/no] | Reason if no | Date of tumor<br>markers<br>sampling | CEA [μg/L] | CA 19-9 [U/L] |
| | | Baseline | | | | | |
| | | Pre-cycle 1 | | | | | |
| | | ••• | | | | | |
| | | Cycle 1 | | | | | |
| | | EOT | | | | | |

# Listing 19: RAS mutation analyses on tumor tissue

| patien<br>t.patie<br>nt_no | registrati<br>on.registr<br>ation_ar<br>m_rando<br>mized | | baselab.basel<br>ab_ras_mutat<br>ion_performe<br>d,<br>precycle.prec<br>ycle_ras_mut<br>ation_perform<br>ed | baselab.baselab _ras_mutation_n d(_spec), precycle.precycle _ras_mutation_n d(_spec) | baselab.ba selab_ras_ mutation_ date, precycle.pr ecycle_ras _mutation _date | baselab.baselab_ras_<br>mutation_m(_spec),<br>baselab.baselab_ras_<br>mutation_m_n(_spec),<br>precycle.precycle_ras_<br>mutation_m(_spec),<br>precycle.precycle_ras_<br>mutation_m_n(_spec) | baselab.base<br>lab_ras_mut<br>ation_status,<br>precycle.prec<br>ycle_ras_mut<br>ation_status | baselab<br>.basela<br>b_kras,<br>precycl<br>e.precy<br>cle_kra<br>s | baselab.bas<br>elab_kras_<br>mutation_list<br>,<br>precycle.pre<br>cycle_kras_<br>mutation_list | baselab<br>.basela<br>b_nras,<br>precycl<br>e.precy<br>cle_nra<br>s | baselab.bas elab_nras_ mutation_list , precycle.pre cycle_nras_ mutation_list |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Patie<br>nt No. | Arm | Poin<br>t in<br>time | RAS mutation<br>analysis on<br>tumor tissue<br>performed<br>[yes/no] | Reason if no | Date of<br>tissue<br>analysis | Method of tissue<br>analysis | RAS mutation status in tissue [wt/mutant] | KRAS<br>detecte<br>d<br>[yes/no] | Exon(s) and<br>Codon(s) of<br>KRAS<br>mutation(s) | NRAS<br>detecte<br>d<br>[yes/no] | Exon(s) and<br>Codon(s) of<br>NRAS<br>mutation(s) |
| | | | Baseline | | | | | | | | |
| | | | Pre-cycle 1 | | | | | | | | |

### Liquid biopsy analyses:

# **Listing 20.1: Samplings for liquid biopsy**

| | registration.registrat<br>ion_arm_randomize<br>d | precycle.p<br>recycle_n<br>o,<br>therapycy<br>cle.therap<br>ycycle_no | baselab.baselab_blood<br>_taken,<br>precycle.precycle_bloo<br>_d_taken,<br>therapycycle.therapycy<br>_cle_blood_taken | baselab.baselab_blo<br>od_nd(_spec),<br>precycle.precycle_bl<br>ood_nd(_spec),<br>therapycycle.therapy<br>cycle_blood_nd(_spe<br>c) | biopsy.biops<br>y_sample_da<br>te | biopsy.biopsy<br>_shipping_dat<br>e | biopsy.biopsy_samp<br>le_analyzed | biopsy.biopsy<br>_sample_ana<br>lyzed_date |
|---|---|---|---|---|---|---|---|---|
| Patient No. | Arm | Point in time | Sampling for liquid biopsy taken [yes/no] | Reason if no | Date of sampling | Date of shipping | Sample intact and analyzable [yes/no] | Date of initial analysis |
| | | Baseline | | | | | | |
| | | Pre-cycle | | | | | | |
| | | 1 | | | | | | |
| | | Cycle 1 | | | | | | |
| | _ | | | | _ | _ | | |

### Listing 20.2: Samplings for liquid biopsy - RAS mutation status

| patient.pa<br>tient_no | registration.registratio<br>n_arm_randomized | biopsy.biopsy_<br>sample_date | biopsy.biopsy_ras_<br>mutation_method | biopsy.biopsy_ras_<br>mutation_status | biopsy.bio<br>psy_kras | biopsy.biopsy_kra<br>s_mutation_list | biopsy.bio<br>psy_nras | biopsy.biopsy_nra<br>s_mutation_list |
|---|---|---|---|---|---|---|---|---|
| Patient<br>No. | Arm | Date of sampling | Method of liquor<br>analysis | RAS mutation<br>status in liquor<br>[wt/mutant] | KRAS<br>detected<br>[yes/no] | Exon(s) and<br>Codon(s) of<br>KRAS mutation(s) | NRAS<br>detected<br>[yes/no] | Exon(s) and<br>Codon(s) of<br>NRAS mutation(s) |

MoLiMoR

EudraCT-No. 2019-003714-14

# Listing 20.3: Samplings for liquid biopsy - first conversion to RASwt

| patient.patie<br>nt_no | registration.registration<br>_arm_randomized | precycle.prec<br>ycle_no | precylce.precyc<br>le_cycle_date | biopsy.biopsy_sample_date | biopsy.biopsy_sa<br>mple_date | |
|---|---|---|---|---|---|---|
| Patient No. | Arm | Point in time | First day of cycle | Date of sampling of liquid biopsy in which conversion to RASwt was detected first | Date of baseline sampling | Time from baseline<br>sampling until first<br>detection of RASwt<br>[days] |
| | | Pre-cycle x | | | | |

# Pregnancy test results:

# Listing 21: β-HCG pregnancy tests

| patient.p<br>atient_no | registr<br>ation.r<br>egistrat<br>ion_ar<br>m_ran<br>domize<br>d | precycle.<br>precycle<br>_no,<br>therapyc<br>ycle.ther<br>apycycle<br>_no | baselab.baselab_preg_test_performed, precycle.precycle_preg_test_performed , therapycycle.therapycycle_preg_test_p erformed, eot.eot_preg_test_performed | baselab.baselab_preg_test_nd(_ | baselab.baselab_preg_<br>test_date,<br>precycle.precycle_preg<br>_test_date,<br>therapycycle.therapycy<br>cle_preg_test_date,<br>eot.eot_date | baselab.baselab_preg_tes |
|---|---|---|---|---|---|---|
| Patient<br>No. | Arm | Point in time | Pregnancy test (urine) performed [yes/no] | Reason if no | Date | Result [positive/negative] |
| | | Baseline | | | | |
| | | Pre-cycle<br>1 | | | | |
| | | Cycle 1 | | | | |
| | | EOT | | | | |

### Treatment cycles:

# Listing 22.1: Treatment cycles - general

| pati<br>ent.<br>pati<br>ent_<br>no | registra<br>tion.reg<br>istratio<br>n_arm_<br>random<br>ized | precycle.precycle_no,<br>therapycycle.therapycycle_no | precycle.precycle _exam_performe d, therapycycle.ther apycycle_exam_ performed | precycle.precycle _exam_reason(_ | precycle.precycle_cyc<br>le_date,<br>therapycycle.therapyc<br>ycle_w1_cycle_date | precycle.precyc<br>le_folfiri_admin,<br>therapycycle.th<br>erapycycle_w1<br>_folfiri_admin | therapycycl<br>e.therapycy<br>cle_surgery<br>_taken | therapy<br>cycle.th<br>erapyc<br>ycle_su<br>rgery_d<br>ate | therap<br>ycycle.<br>therap<br>ycycle<br>_surge<br>ry_type |
|---|---|---|---|---|---|---|---|---|---|
| Pati<br>ent<br>No. | Arm | Point in time | Examinations<br>and/or treatment<br>performed<br>[yes/no] | Reason if no | First day of cycle | Study<br>treatment<br>administered<br>[yes/no] | Resection of<br>metastases<br>since last<br>visit [yes/no] | Date of surgery | Resect<br>ed<br>metast<br>ases |
| | | Pre-cycle 1 | | | | | | | |
| | | ••• | | | | | | | |
| | | Cycle 1 | | | | | | | |
| | | ••• | | | | | | | |

# Listing 22.2: Treatment cycles - irinotecan (iv infusion, 180 mg/m² over 30-90 min)

| pati<br>ent. | regist<br>ration<br>.regist<br>ration | precycle.precycle_no,<br>therapycycle.therapyc<br>ycle_no, | precycle.prec<br>ycle_irino_ad<br>min, | precycle.pre<br>cycle_irino_<br>nd(_spec), | precycle.pre<br>cycle_irino_<br>batch, | precycle.precycl<br>e_irino_admin_<br>date(_nd), | precycle.pr<br>ecycle_irino<br>_pro, | precycle.precyc<br>le_irino_pro_nd<br>(_spec), | precycle.prec<br>ycle_irino_du<br>ration, | precycle.pre<br>cycle_irino_<br>dose, |
|---|---|---|---|---|---|---|---|---|---|---|
| pati<br>ent_<br>no | _arm<br>_rand<br>omize<br>d | therapycycle.therapyc<br>ycle_w1_cycle_no,<br>therapycycle.therapyc<br>ycle_w2_cycle_no | therapycycle.t<br>herapycycle_i<br>rino_admin | therapycycle<br>.therapycycl<br>e_irino_nd(_<br>spec) | therapycycle<br>.therapycycl<br>e_irino_batc<br>h | therapycycle.the<br>rapycycle_irino_<br>admin_date(_nd<br>) | therapycycl<br>e.therapycy<br>cle_irino_pr<br>o | therapycycle.th<br>erapycycle_irin<br>o_pro_nd(_spe<br>c) | therapycycle.<br>therapycycle<br>_irino_durati<br>on | therapycycl<br>e.therapycy<br>cle_irino_do<br>se |
| | | | Irinotecan | | | | Prolonged | | lf | |
| Pati<br>ent<br>No. | Arm | Point in time | administered<br>in standard<br>dose [yes/no] | Reason if no | Batch | Date | infusion<br>duration<br>[yes/no] | Reason if yes | Infusion<br>duration<br>[min] | Dose<br>[mg/m²] |
| ent | Arm | Point in time Pre-cycle 1 | administered<br>in standard | Reason if no | Batch | Date | infusion<br>duration | Reason if yes | duration | |
| ent | Arm | | administered<br>in standard | Reason if no | Batch | Date | infusion<br>duration | Reason if yes | duration | |
| ent | Arm | Pre-cycle 1 | administered<br>in standard | Reason if no | Batch | Date | infusion<br>duration | Reason if yes | duration | |

# Listing 22.3: Treatment cycles - folinic acid (iv infusion, 400 mg/m² over 120 min)

| pati<br>ent.<br>pati<br>ent_<br>no | regist ration regist ration arm rand omize d | precycle.precycle_no,<br>therapycycle.therapyc<br>ycle_no,<br>therapycycle.therapyc<br>ycle_w1_cycle_no,<br>therapycycle.therapyc<br>ycle_w2_cycle_no | n, | precycle.prec<br>ycle_fa_admi<br>n_nd(_spec),<br>therapycycle.t<br>herapycycle_f<br>a_admin_nd(<br>spec) | precycle.pr<br>ecycle_fa_<br>batch,<br>therapycycl<br>e.therapycy<br>cle_fa_batc<br>h | precycle.precyc le_fa_admin_d ate(_nd), therapycycle.th erapycycle_fa_ admin_date(_n d) | precycle.pre<br>cycle_fa_pr<br>olong,<br>therapycycle<br>.therapycycl<br>e_fa_prolon<br>g | precycle.precycl e_fa_prolong_n d(_spec), therapycycle.the rapycycle_fa_pr olong_nd(_spec ) | cycle_fa_dur<br>ation,<br>therapycycle | precycle.pr<br>ecycle_fa_<br>dose,<br>therapycycl<br>e.therapycy<br>cle_fa_dos<br>e |
|---|---|---|---|---|---|---|---|---|---|---|
| Pati<br>ent<br>No. | Arm | Point in time | Folinic acid<br>administered<br>in standard<br>dose [yes/no] | Reason if no | Batch | Date | Prolonged infusion duration [yes/no] | Reason if yes | Infusion<br>duration<br>[min] | Dose<br>[mg/m²] |
| | | Pre-cycle 1 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | Cycle 1 | | · | | · | | <u>-</u> | _ | |
| | | ••• | | | | | | | | |

### Listing 22.4: Treatment cycles - 5-FU (bolus, 400 mg/m²)

| pati<br>ent.<br>pati<br>ent_<br>no | registra<br>tion.reg<br>istratio<br>n_arm_<br>random<br>ized | precycle.precycle_no, therapycycle.therapycycle_w1_cycle_no, therapycycle.therapycycle_w2_cycle_no | precycle.precycle<br>_ffu1_admin,<br>therapycycle.ther<br>apycycle_ffu1_a<br>dmin | precycle.precycle_ff u1_admin_nd(_spec ), therapycycle.therapy cycle_ffu1_admin_n d(_spec) | | precycle.precycle_ffu1_<br>admin_date(_nd),<br>therapycycle.therapycyc<br>le_ffu1_admin_date(_n<br>d) | precycle.pre<br>cycle_<br>ffu1_dose,<br>therapycycle.<br>therapycycle<br>_ ffu1_dose |
|---|---|---|---|---|---|---|---|
| Pati<br>ent<br>No. | Arm | Point in time | 5-FU bolus<br>administered in<br>standard dose<br>[yes/no] | Reason if no | Batch | Date | Dose<br>[mg/m²] |
| | | Pre-cycle 1 | | | | | |
| | | ••• | | | | | |
| | | Cycle 1 | | | | | |
# Listing 22.5: Treatment cycles - 5-FU (iv infusion, 2400 mg/m² over 46 h)

| pati<br>ent.<br>pati<br>ent_<br>no | registra<br>tion.reg<br>istratio<br>n_arm_<br>random<br>ized | precycle.precycle_no, therapycycle.therapycycle _no, therapycycle.therapycycle _w1_cycle_no, therapycycle.therapycycle _w2_cycle_no | precycle.precy<br>cle_ffu2_admi<br>n,<br>therapycycle.t<br>herapycycle_<br>ffu2_admin | precycle.prec ycle_ffu2_ad min_nd(_spec ), therapycycle.t herapycycle_f fu2_admin_n d(_spec) | precycle.p<br>recycle_ff<br>u2_batch,<br>therapycy<br>cle.therap<br>ycycle_ffu<br>2_batch | precycle.pre cycle_ffu2_a dmin_date(_ nd), therapycycle .therapycycl e_ffu2_admi n_date(_nd) | precycle.pre<br>cycle_ffu2_p<br>rolong,<br>therapycycle<br>.therapycycl<br>e_ffu2_prolo<br>ng | precycle.pre cycle_ffu2_p rolong_nd(_ spe), therapycycle .therapycycl e_ffu2_prolo ng_nd(_spe) | precycle.pre<br>cycle_ffu2_d<br>uration,<br>therapycycle<br>.therapycycl<br>e_ffu2_durat<br>ion | precycle.pre<br>cycle_ffu2_d<br>ose,<br>therapycycle<br>.therapycycl<br>e_ffu2_dose |
|---|---|---|---|---|---|---|---|---|---|---|
| Pati<br>ent<br>No. | Arm | Point in time | 5-FU infusion<br>administered<br>in standard<br>dose [yes/no] | Reason if no | Batch | Date | Prolonged<br>infusion<br>duration<br>[yes/no] | Reason if yes | Infusion<br>duration<br>[min] | Dose<br>[mg/m²] |
| | | Pre-cycle 1 | | | | | | | | |
| | | Cycle 1 | | | | | | | | |
| | | ••• | | | | | | | | |

### Listing 22.6: Treatment cycles - cetuximab (iv infusion, initially 400mg/m<sup>2</sup> over 120 min, subsequently 250 mg/m<sup>2</sup> over 60 min)

| patie<br>nt.pa | registr<br>ation.r<br>egistra<br>tion ar | therapycycle.th | therapycycle.therapycy<br>cle_w1_ce_admin, | therapycycle.t<br>herapycycle_<br>w1_ce_nd(_s<br>pec), | therapycycl<br>e.therapycy<br>cle_w1_ce<br>_batch, | therapycycle.t<br>herapycycle_w<br>1_ce_admin_d<br>ate(_nd), | therapycyc<br>le.therapy<br>cycle_w1_<br>ce_pro, | therapycycle.t<br>herapycycle_<br>w1_ce_pro_n<br>d(_spec), | therapycycle.<br>therapycycle<br>_w1_ce_od_<br>duration, | therapycycl<br>e.therapycy<br>cle_w1_ce(<br>_od)_dose, |
|---|---|---|---|---|---|---|---|---|---|---|
| tient<br>_no | m_ran<br>domize<br>d | erapycycle_no | therapycycle.therapycy cle_w2_ce_infu_admin | therapycycle.t<br>herapycycle_<br>w2_ce_infu_n<br>d(_spec) | therapycycl<br>e.therapycy<br>cle_w2_ce<br>_batch | therapycycle.t<br>herapycycle_w<br>2_ce_admin_d<br>ate(_nd) | therapycyc<br>le.therapy<br>cycle_w2_<br>ce_pro | therapycycle.t<br>herapycycle_<br>w2_ce_pro_n<br>d(_spec) | therapycycle.<br>therapycycle<br>_w2_ce_od_<br>duration | therapycycl<br>e.therapycy<br>cle_w2_ce_<br>od_dose |
| Pati<br>ent<br>No. | Arm | Point in time | Cetuximab<br>administered in<br>standard dose [yes/no] | Reason if no | Batch | Date | Prolonged infusion duration [yes/no] | Reason if yes | Infusion<br>duration<br>[min] | Dose<br>[mg/m²] |
| | | Cycle 1 week 1 | | | | | | | | |
| | | Cycle 1 week 2 | | | | | · | | | |

### Primary and secondary objectives:

# Listing 23.1: RECIST assessments

| patie<br>nt.p<br>atien<br>t_no | registr<br>ation.r<br>egistr<br>ation_<br>arm_r<br>ando<br>mized | precycle<br>.precycl<br>e_no,<br>therapyc<br>ycle.ther<br>apycycle<br>_no | baseline.baseline_rec<br>ist_tm_performed,<br>precycle.precycle_rec<br>ist_tm_performed,<br>therapycycle.therapyc<br>ycle_recist_tm_perfor<br>med | 2d00iii10:2d00iii10_100i0t_tii1_1id(_0p0d0); | tm_s<br>t.tm<br>_st_<br>st_n<br>r | | tm.tm_loc_<br>metastasis<br>_count | tm_st.<br>tm_st<br>_mea<br>s_am<br>ount | tm_<br>st.t<br>m_s<br>t_tot<br>al | tm_st.tm_st_c<br>onsultations | Tm _st.t m_s t_co mm ent |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Pati<br>ent<br>No. | Arm | Point in time | RECIST assessment performed [yes/no] | Reason | Stag<br>ing<br>No. | Date of<br>RECIS<br>T<br>assess<br>ment | Number of<br>metastase<br>s at<br>beginning<br>of the<br>study | Sum<br>of<br>sizes<br>[mm] | Ove<br>rall<br>ass<br>ess<br>men<br>t | Consultation with Administratio n Office has occurred [yes/no] | Co<br>mm<br>ent |
| | | Baseline | | | | | _ | | | | |
| | | Pre- | | | | | | | | | |
| | | cycle 1 | | | | | | | | | |
| | | Cycle 1 | | | | | | | | | |

# Listing 23.2: RECIST assessments - lesions

| patient.p<br>atient_no | registration.registratio<br>n_arm_randomized | tm_st.tm<br>_st_st_nr | tm_st.tm<br>_st_date | tm_le.tm<br>_le_loc | tm_le.tm_l<br>e_loc_ext | tm_le.tm_l<br>e_method | tm_le.tm<br>_le_size | tm_le.tm_le_<br>tumor_type | tm_st.tm_st_mea<br>s_assessment | tm_st.tm_st_imme<br>as_assessment |
|---|---|---|---|---|---|---|---|---|---|---|
| Patient<br>No. | Arm | Staging<br>No. | Date | Localiza<br>tion | Detailed<br>informatio<br>n about<br>localizatio<br>n | Method | Size of<br>lesion if<br>measura<br>ble [mm] | Tumor type if<br>non-<br>measurable | Assessment<br>measurable<br>lesions | Assessment non-<br>measurable<br>lesions |

# Listing 24: PFS, OS, and TFTS

| | omized Stored_at | _contact_date | | ae.ae_ffu_inter_date,<br>ae.ae_ce_inter_date | | m_st_d<br>ate | | y_death_d<br>ate | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient Arı | Arm Date of randomization | Date of last<br>contact | Treatment<br>discontinuation<br>for any reason<br>[yes/no] | Date of (first)<br>discontinuation | Progr<br>ession<br>[yes/n<br>o] | Date of progres sion | Death<br>[yes/no] | Date of<br>death | PFS<br>[mo<br>nths<br>] | OS<br>[mo<br>nths<br>] | TFT<br>S<br>[mo<br>nths<br>] |

### End of treatment:

# Listing 25.1: EOT - resection and new therapy

| patient.p<br>atient_no | registration.registratio<br>n_arm_randomized | eot.eot<br>_date | eot.eot_end_reaso<br>n(_other_spec) | eot.eot_resecti<br>on_date | eot.eot_resection<br>_status | eot.eot_tumor_th | tumor.tum<br>or_therapy | tumor.tum<br>or_start | tumor.tumor<br>_end(_nd) |
|---|---|---|---|---|---|---|---|---|---|
| Patient<br>No. | Arm | EOT<br>evaluati<br>on date | Reason for EOT | Resection date if resection performed | Resection status if resection performed | New tumor<br>therapy since last<br>study treatment<br>[yes/no] | New<br>therapy | Start date<br>of new<br>therapy | End date of new therapy |
| | | | | · | | | | | |

# Listing 25.2: EOT - RAS mutation status

| patient.p<br>atient_no | registration.registrati<br>on_arm_randomize<br>d | eot.eot_ras_mutation_st<br>atus_done | eot.eot_ras_mu<br>tation_status | eot.eot_kras | eot.eot_kras_mutatio<br>n_list | eot.eot_nras | eot.eot_nras_mutation<br>_list |
|---|---|---|---|---|---|---|---|
| Patient | ۸۳۳۰ | Results of RAS mutation | Mutation status | KRAS detected | Exon(s) and Codon(s) | NRAS detected | Exon(s) and Codon(s) |
| No. | Arm | status available [yes/no] | [wt/mutant] | [yes/no] | of KRAS mutation(s) | [yes/no] | of NRAS mutation(s) |

# Follow-up visits:

### Listing 26.1: Follow-up visit - first part

| | registration.registration_arm_randomized | | | followup.follo<br>wup_contact | followup_tumor_th | tumor.tumo<br>r_therapy | tumor.tumor_<br>start | tumor.tumor_e<br>nd(_nd) |
|---|---|---|---|---|---|---|---|---|
| Patient No. | Arm | Follow-up<br>No. | Follow-up visit<br>date | Contact with patient | Changes in new therapy since last visit [yes/no] | New<br>therapy | Start date of<br>new therapy | End date of new therapy |

# Listing 26.2: Follow-up visit - second part

| | registration.registrati<br>on_arm_randomized | | followup_followup_surgery_taken | followup_followup_s<br>urgery_date | followup_followup_surgery_type |
|---|---|---|---|---|---|
| Patient No. | Arm | Follow-up No. | Resection of metastases since last visit [yes/no] | Date of resection | Which metastasis were resected |

### End of study:

# Listing 27: End of study

| I Arm I | Reason for<br>end of study | Date of<br>death if<br>applicable | Reason of<br>death if<br>applicable | nci_v5_a<br>e.ae | <br>Death related<br>disease if<br>applicable | Date of<br>withdrawal if<br>applicable | Reason of<br>withdrawal if<br>applicable |
|---|---|---|---|---|---|---|---|

### Adverse events:

Listing 28.1: AEs/toxicity - terminology, timeline, and causality

| patient.pa<br>tient_no | registration.registration<br>_arm_randomized | | ae.ae_st<br>art(_na) | ae.ae_e<br>nd(_na) | ae.ae_o<br>utcome | ae.ae_treatm<br>ent_started | | ae.ae_irino _causal, ae.ae_fa_c ausal, ae.ae_ffu_ causal, ae.ae_ce_ causal | ae.ae_irin o_action, ae.ae_fa_ action, ae.ae_ffu_ action, ae.ae_ce_ action | ae.ae_medicat<br>ion_treated |
|---|---|---|---|---|---|---|---|---|---|---|
| Patient<br>No. | Arm | Terminology a to CTCAE ve ae.a nci_v5 e_nci _ae.ae Grad e Term | Start<br>date | End date | Outcom<br>e | Study<br>treatment<br>started<br>[yes/no] | Study<br>treat<br>ment<br>comp<br>onent | Causal<br>relationshi<br>p<br>suspected<br>[yes/no] | Action<br>taken | Event treated<br>with<br>medication<br>[yes/no] |

# Listing 28.2: AEs/toxicity - SAEs and special AEs

| Patient No. Arm ae.a v5_ e_n Start date [yes/no] serious [yes/no] | patient.patie<br>nt_no | registrati<br>on.regist<br>ration_ar<br>m_rando<br>mized | ae.ae_start(_na | ae.ae_sae | ae.ae_criteria_fatal, ae.ae_criteria_life_threatening, ae.ae_criteria_hospital, ae.ae_criteria_disability, ae.ae_criteria_congenital, ae.ae_criteria_important_event (_spec) | ae.ae_special | ae.ae_criteria_pregnancy,<br>ae.ae_criteria_error |
|---|---|---|---|---|---|---|---|
| Gra Ter Oth de m er | Patient No. | Arm | according to CTCAE version 5 ae.a | | _ | | Reason for classification as special |

### 5.3 Figures

Figure 1: Swimmer plot



Figure 2: Progression-free survival (PFS) [months]

| Figure | Figure 2 | Example (no study data) |
|---|---|---|
| Title 1 | Progression-free survival (PFS) [months] | 1.0 |
| Title 2 | | 0.9 |
| Type of graph | Kaplan-Meier plot | + |
| y-axis | 0 to 1 | 0.8 |
| y-axis (label) | PFS | 0.7 |
| x-axis | 0 to maximum event time | 0.6 |
| x-axis (label) | Months | <u>ω</u> 0.5 |
| Legend | Study arms A and B and Total | 0.4 |
| Footnote | | |
| Additional | Patients at risk will be displayed for specified | 0.3 |
| information | timepoints on x-axis. One PFS curve for each study arm and the total population will be | 0.2 |
| | displayed. Due to the small number of patients, no p-value will be displayed. | 0.1 |
| | no p-value will be displayed. | 0.0 + Censored |
| | | A 11 10 9 8 5 4 1 1 1<br>B 11 10 10 9 7 5 3 |
| | | Total 22 20 19 17 12 9 4 1 0 1 2 3 4 5 6 7 |
| | | Months |
| | | ARM — A — B — Total |

Figure 3: Overall survival (OS) [months]

| Figure | Figure 3 | Example (no study data, no matching y-axis label) |
|---|---|---|
| Title 1 | Overall survival (OS) [months] | 1.0 |
| Title 2 | | |
| Type of graph | Kaplan-Meier plot | 0.9 |
| y-axis | 0 to 1 | 0.8 |
| y-axis (label) | os | 0.7 |
| x-axis | 0 to maximum event time | 0.6 |
| x-axis (label) | Months | ω 0.5 |
| Legend | Study arms A and B and Total | 0.4 |
| Footnote | | |
| Additional | Patients at risk will be displayed for specified | 0.3 |
| information | timepoints on x-axis. One OS curve for each study arm and the total population will be | 0.2 |
| | displayed. Due to the small number of patients, no p-value will be displayed. | 0.1 |
| | no p-value will be displayed. | 0.0 - + Censored |
| | | A 11 10 9 8 5 4 1 1 1 B 11 10 10 9 7 5 3 |
| | | Total 22 20 19 17 12 9 4 1 1 0 1 2 3 4 5 6 7 |
| | | Months |
| | | ARM ———————————————————————————————————— |

Figure 4: Time to failure of treatment strategy (TFTS) [months]

| Figure | Figure 4 | Example (no study data, no matching y-axis label) |
|---|---|---|
| Title 1 | Time to failure of treatment strategy (TFTS) [months] | 1.0 |
| Title 2 | | 0.9 |
| Type of graph | Kaplan-Meier plot | 0.8 |
| y-axis | 0 to 1 | 0.7 |
| y-axis (label) | TFTS | 0.6 |
| x-axis | 0 to maximum event time | |
| x-axis (label) | Months | <u>V</u> 0.5 |
| Legend | Study arms A and B and Total | 0.4 |
| Footnote | | 0.3 |
| Additional information | Patients at risk will be displayed for specified timepoints on x-axis. One TFTS curve for each study arm and the total population will be displayed. Due to the small number of patients, | 0.2 |
| | no p-value will be displayed. | 0.0 + Censored A 11 10 9 8 5 4 1 1 |
| | | A 11 10 9 8 5 4 1 1 1 B 10 10 9 7 5 3 Total 22 20 19 17 12 9 4 1 |
| | | 0 1 2 3 4 5 6 7 Months |
| | | ARM — A B — Total |

#### 6 Statistical software

All descriptive statistical analyses will be performed by using the statistical software SAS version 9.4.

#### 7 Medical dictionaries

As medical dictionary for analysis we use the latest available version of MedDRA and ICD10.

#### 8 Coding conventions

There are no special coding conventions.

#### 9 Output format

If a statistical report will be written, the respective tables and figures will be presented in the text. The text will be written in Arial 11 pt with 1.0 line spacing with exceptions to title and signature pages. The TLF will be written in Arial 10 pt and dates contained in TLF will be given in DDMMMYY format.

#### 10 List of the tables, listings, and figures planned for the Final Statistical Report

### Tables:

- Table 1: General data
- Table 2: Patients' first conversion to RAS wild-type
- Table 3: Patient responses
- (Optionally) Table 4.1: AEs overview
- (Optionally) Table 4.2: AEs System Organ Class (SOC) and Preferred Term (PT) by NCI CTCAE grade
- (Optionally) Table 4.3: AEs number of patients with respect to System Organ Class (SOC) and Preferred Term (PT) by maximal NCI CTCAE grade

#### Listings:

- Listing 1.1: Inclusion criteria
- Listing 1.2: Inclusion criteria 01-09
- Listing 1.3: Inclusion criteria 10-19
- Listing 2.1: Exclusion criteria
- Listing 2.2: Exclusion criteria 01-08
- Listing 2.3: Exclusion criteria 09-15
- Listing 2.4: Exclusion criteria 16-22
- Listing 3: Eligibility, enrollment, and randomization
- Listing 4: Patient demographics
- Listing 5.1: Initial diagnosis of mCRC TNM staging
- Listing 5.2: Initial diagnosis of mCRC resection
- Listing 5.3: Initial diagnosis of mCRC RAS mutation analysis
- Listing 6: Medical history
- Listing 7.1: Relevant medication premedication
- Listing 7.2: Relevant medication concomitant medication
- Listing 8: Baseline echocardiography
- Listing 9: Baseline TNM staging
- Listing 10: Baseline coagulation parameters
- Listing 11: Baseline DPD deficiency
- Listing 12: Baseline hepatitis serology
- Listing 13: ECG assessments
- Listing 14: ECOG performance statuses

- Listing 15: Vital signs
- Listing 16: Hematological lab assessments
- Listing 17.1: Blood chemistry lab assessments first part
- Listing 17.2: Blood chemistry lab assessments second part
- Listing 18: Tumor markers lab assessments
- Listing 19: RAS mutation analyses on tumor tissue
- Listing 20.1: Samplings for liquid biopsy
- Listing 20.2: Samplings for liquid biopsy RAS mutation status
- Listing 20.3: Samplings for liquid biopsy first conversion to RASwt
- Listing 21: β-HCG pregnancy tests
- Listing 22.1: Treatment cycles general
- Listing 22.2: Treatment cycles irinotecan (iv infusion, 180mg/m<sup>2</sup> over 90 min)
- Listing 22.3: Treatment cycles folinic acid (iv infusion, 400mg/m<sup>2</sup> over 120 min)
- Listing 22.4: Treatment cycles 5-FU (bolus, 400mg/m²)
- Listing 22.5: Treatment cycles 5-FU (iv infusion, 2400mg/m² over 46h)
- Listing 22.6: Treatment cycles cetuximab (iv infusion, initially 400 mg/m² over 120 min, subsequently 250 mg/m² over 60 min)
- Listing 23.1: RECIST assessments
- Listing 23.2: RECIST assessments lesions
- Listing 24: PFS, OS, and TFTS
- Listing 25.1: EOT resection and new therapy
- Listing 25.2: EOT RAS mutation status
- Listing 26.1: Follow-up visit first part
- Listing 26.2: Follow-up visit second part
- Listing 27: End of study
- Listing 28.1: AEs/toxicity terminology, timeline, and causality
- Listing 28.2: AEs/toxicity SAEs and special AEs

#### Figures:

- Figure 1: Swimmer plot
- Figure 2: Progression-free survival (PFS) [months]
- Figure 3: Overall survival (OS) [months]
- Figure 4: Time to failure of treatment strategy (TFTS) [months]

# 11 History table

| Version | Version of Mock-ups | Date<br>[DDMMMYY] | Author | Sections changed | Brief description of change |
|---|---|---|---|---|---|
| Draft<br>v0.1 | First version | 18FEB22 | Dr. Maximilian<br>Parr | None | First version, hence no changes |
| Draft<br>v0.2 | Second version | 11MAR22 | Dr. Maximilian<br>Parr | Title pages | Actualized |
| | | | | Section 4.12 | Added some conventions |
| | | | | Chapter 5 | Mostly minor adjustments to tables and listings |
| Draft<br>v0.3 | Third version | 18MAR22 | Dr. Maximilian<br>Parr | Chapter 5 | A few more minor changes in listings |
| Draft<br>v0.4 | Fourth<br>version | 31MAR22 | Dr. Maximilian<br>Parr | Section 4.12 | Added time conventions |
| | | | | Chapter 5 | Added third table and Listing 20.3 |
| | | 14APR22 | Dr. Maximilian<br>Parr | Section 4.3.9,<br>Section 5.1,<br>Section 10 | Added optionally tables for AEs and their references |
| | | 23NOV22 | Dr. Maximilian<br>Parr | Section 4.12 | Spelling mistake |
| | | 06MAR23 | Dr. Maximilian<br>Parr | overall | Typos and preparation of Version 1.0 |
| Version<br>0.9 | Pre-final version | 16MAR23 | Dr. Maximilian<br>Parr | overall | Typos and overseen changes |
| Version<br>1.0 | Final<br>version | 06JUN23 | Dr. Maximilian<br>Parr | overall | Incorporating pre-final review feedback |
| | | 22JUN23 | Dr. Maximilian<br>Parr | Section 4.12,<br>Section 4.17 | Wording and typo |
| Version<br>2.0 | Final<br>Version | 12SEP24 | Dr. Maximilian<br>Parr | Section 4.2,<br>4.3.5, and<br>4.3.6 | Added parts for graphical Kaplan-Meier for PFS, OS, and TFTS |
| | | | | Section 5.3 and 10 | Added three figures |